CLINICAL TRIAL: NCT01983592
Title: An N-of-1 Study of Homeopathic Treatment of Fatigue in Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Canadian CAM Research Fund (Unknown); Ottawa Integrative Cancer Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 194318
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Fatigue; Effects of Chemotherapy
Keywords: Homeopathy; Fatigue; Chemotherapy; Cancer
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homeopathic medicine (Active Comparator): The study medication will be administered in one of two forms: (1) 3.5 mm diameter lactose/sucrose globule to be administered sublingually; or (2) 3.5 mm diameter lactose/sucrose globule dissolved in 250 ml spring water and administered orally. The medication will be administered as either 1 globule sublingual or 5 mL oral remedy/water up to 3 times per day. The dosage regimen is varialble at the discretion of the study clinician.
  Interventions: Other: Homeopathic medicine
- Unmedicated lactose/sucrose globule (Placebo Comparator): The placebo will be administered in one of two forms: (1) 3.5 mm diameter lactose/sucrose globule to be administered sublingually; or (2) 3.5 mm diameter lactose/sucrose globule dissolved in 250 ml spring water and administered orally. The medication will be administered as either 1 globule sublingual or 5 mL oral remedy/water up to 3 times per day. The dosage regimen is varialble at the discretion of the study clinician.
  Interventions: Other: Unmedicated lactose/sucrose globule

INTERVENTIONS:
Other: Homeopathic medicine — Intervention must begin within 5 days of chemotherapy cycle completion. Intervention will continue until the next cycle of chemotherapy. The initial consultation will involve a verbal interview between the homeopath and the participant. The practitioner will then choose a single homeopathic remedy that will focus on the reduction of fatigue. Only one homeopathic remedy and potency will be administered at a given time. The participant will be asked to take the study medication at least 30 minutes before or after taking other medications, food and strong smelling substances.
  Arms: Homeopathic medicine
Other: Unmedicated lactose/sucrose globule
  Arms: Unmedicated lactose/sucrose globule

SUMMARY:
Fatigue is frequently identified as one of the most troublesome symptoms in cancer patients and there are very few conventional therapies which can address the symptom of fatigue in patients who are undergoing cancer treatment.

This study will be testing whether the administration of a complementary therapy (individualized homeopathy) to a patient undergoing chemotherapy treatment is feasible and whether this treatment can lessen the fatigue symptoms of adults. The study will also test whether the n-of-1 study design is feasible in this population.

DETAILED DESCRIPTION:
This is an n-of-1 pilot trial of individualized homeopathic treatment of fatigue in a single adult who is undergoing any type of chemotherapy administered intermittently (i.e. not continuously). The participant will have a homeopathic consultation within 3 days of a round of chemotherapy ("treatment period") and will be administered either verum or placebo according to a binary randomization allocation sequence unknown to both the clinician and participant. During the subsequent treatment period the participant will be given the other allocation (verum or placebo). The following pairs of allocations will also be randomized with treatment continuing for as long as the participant is undergoing chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of cancer. Patient may have newly diagnosed, relapsed or a second malignant disease.
* Receiving any type of cytotoxic chemotherapy with 6 or more cycles post study enrollment administered intermittently every two or three weeks with no planned radiation treatment.
* Is experiencing fatigue due to the chemotherapy treatments. (or has a score of 2 or higher on the fatigue item of the Symptom Distress Scale)
* Above 18 years of age.
* Able to ingest medications in lactose/sucrose globule or liquid form.

Exclusion Criteria:

* Previous history of allergy to the homeopathic products.
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) | 7 days
  The Multidimensional Fatigue Inventory (MFI) is a 20-item, multi-dimensional, self-report instrument designed to measure fatigue. It covers the following 5 dimensions: 1) General Fatigue, 2) Physical Fatigue, 3) Mental Fatigue, 4) Reduced Motivation and 5) Reduced Activity.

SECONDARY OUTCOMES:
EORTC-QLQ-C30 | 7 days
  The EORTC QLQ-C30 is a 30-item multi-dimensional questionnaire developed to assess the quality of life of cancer patients in the following four domains: functional scales; symptom scales; global quality of life; and single items.

CONTACTS AND LOCATIONS:
Overall Officials: Dugald Seely, ND, Principal Investigator — Canadian College of Naturopathic Medicine
Locations (1):
- Ottawa Integrative Cancer Centre, Ottawa, Ontario, Canada